CLINICAL TRIAL: NCT05506319
Title: Incidence of Hypotension in the Weaning From Vasopressor Drugs
Brief Title: Hypotension in the Weaning From Vasopressor Drugs
Acronym: RENOVA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Nossa Senhora da Conceicao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 57213022.0.0000.5530
Record Dates: First submitted 2022-07-25; First posted 2022-08-18 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Septic Shock
Keywords: vasoconstrictor agents; sepsis; critical care; vasopressin
MeSH Terms: conditions — Shock, Septic; Sepsis; Diabetes Insipidus | interventions — Norepinephrine; Vasopressins

STUDY DESIGN:
Intervention Model Description: A randomized, parallel, open-case clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- norepinephrine group (Experimental): Initial suspension of norepinephrine.
  Interventions: Other: Norepinephrine
- vasopressin group (Experimental): Initial suspension of vasopressin.
  Interventions: Other: Vasopressin

INTERVENTIONS:
Other: Norepinephrine — The patients will be randomized for the initial suspension of norepinephrine (norepinephrine group).
  Arms: norepinephrine group
Other: Vasopressin — The patients will be randomized for the initial suspension of vasopressin (vasopressin group).
  Arms: vasopressin group

SUMMARY:
Although there is consensus in the literature on hemodynamic management of septic shock in the resuscitation phase, the best way to conduct the weaning of vasopressor drugs in the stabilization phase remains open. The present study aims to study the incidence of hypotension in the weaning phase of vasopressor drugs- norepinephrine and vasopressin.

DETAILED DESCRIPTION:
A randomized, open-case clinical trial with 2 arms will be conducted: initial suspension of norepinephrine (norepinephrine group) versus initial vasopressin (vasopressin group).

The selection of patients who will participate in the study will be for convenience. The randomization of the patients will be done by opaque envelopes 1:1, grouped into blocks, generated by random numbers.

The study will be carried out in the intensive care unit of a tertiary hospital in Southern Brazil, taking into account the clinical and surgical patients. In the intensive care unit, after randomization, patients will be identified by posters, attached to the bed. The titration of vasoactive drugs will be criterion of the assistant team.

ELIGIBILITY:
Inclusion Criteria:

* Patients with septic shock, according to the definitions of SEPSIS - 3: septic and hypotensive patients, demanding use of vasoactive drug and lactate greater than 2 mmol/L (18 mg/dL).
* Patients admitted to the intensive care unit.
* Patients in need of associated use of norepinephrine and vasopressin.

Exclusion Criteria:

* Patients in whom discontinuation of norepinephrine or vasopressin has been given by decision of the assistant team, from a perspective of prioritizing palliative care.
* Patients using a combination of a third drug, with the effect of predominantly vasopressor - adrenaline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of hypotension | The first 24 hours after the start of reduction of one of the vasopressors.
  Evaluation of the incidence of hypotension in the first 24 hours after discontinuation of one of the vasoactive drugs: norepinephrine or vasopressin. It is defined as hypotension the drop in mean blood pressure below 65 mmHg, triggering one or more of the following measures: a) administration of crystalloid or colloid aliquot, b) dose increase of the remaining vasoactive drug or c) re-establishment of the drug vasoactive paused.

SECONDARY OUTCOMES:
Mortality | Mortality in a 28-day follow-up, from the beginning of the reduction of one of the vasopressors.
  Evaluation of the mortality in first 28 days after discontinuation of one of the vasoactive drugs.
Length of stay in intensive care unit | In a 28-day follow-up, from the beginning of reduction of one of the vasopressors.
  Evaluation of the length of stay in intensive care unit.
Time of use of the vasoactive drugs | Follow-up of up to 7 days, from the beginning of reduction of one of the vasopressors.
  Quantify the time spent using vasoactive drugs after the removal of the first drug (norepinephrine or vasopressin) in days.
Incidence of arrhythmias | The first 24 hours after the start of reduction of one of the vasopressors.
  Quantify the incidence of arrhythmias with hemodynamic repercussions in 24 hours after withdrawal of the first drug (norepinephrine or vasopressin). This group includes events in which hemodynamic worsening required electrical or chemical cardioversion.
Incidence of hemodialysis | The first 72 hours after the start of reduction of one of the vasopressors.
  Quantify the incidence of hemodialysis, independent of dialysis modality, excluding patients on dialysis chronic.

CONTACTS AND LOCATIONS:
Overall Officials: Cassio Mallmann, MD, Principal Investigator — casmallmann@yahoo.com.br
Locations (1):
- Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Landry DW, Oliver JA. The pathogenesis of vasodilatory shock. N Engl J Med. 2001 Aug 23;345(8):588-95. doi: 10.1056/NEJMra002709. No abstract available. PMID 11529214
- [Result] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Hylander Moller M, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock 2021. Crit Care Med. 2021 Nov 1;49(11):e1063-e1143. doi: 10.1097/CCM.0000000000005337. No abstract available. PMID 34605781
- [Result] Russell JA, Walley KR, Singer J, Gordon AC, Hebert PC, Cooper DJ, Holmes CL, Mehta S, Granton JT, Storms MM, Cook DJ, Presneill JJ, Ayers D; VASST Investigators. Vasopressin versus norepinephrine infusion in patients with septic shock. N Engl J Med. 2008 Feb 28;358(9):877-87. doi: 10.1056/NEJMoa067373. PMID 18305265
- [Result] Der-Nigoghossian C, Hammond DA, Ammar MA. Narrative Review of Controversies Involving Vasopressin Use in Septic Shock and Practical Considerations. Ann Pharmacother. 2020 Jul;54(7):706-714. doi: 10.1177/1060028020901521. Epub 2020 Jan 20. PMID 31958982
- [Result] Russell JA, Fjell C, Hsu JL, Lee T, Boyd J, Thair S, Singer J, Patterson AJ, Walley KR. Vasopressin compared with norepinephrine augments the decline of plasma cytokine levels in septic shock. Am J Respir Crit Care Med. 2013 Aug 1;188(3):356-64. doi: 10.1164/rccm.201302-0355OC. PMID 23796235
- [Result] Gordon AC, Wang N, Walley KR, Ashby D, Russell JA. The cardiopulmonary effects of vasopressin compared with norepinephrine in septic shock. Chest. 2012 Sep;142(3):593-605. doi: 10.1378/chest.11-2604. PMID 22518026
- [Result] Nascente APM, Freitas FGR, Bakker J, Bafi AT, Ladeira RT, Azevedo LCP, Lima A, Machado FR. Microcirculation improvement after short-term infusion of vasopressin in septic shock is dependent on noradrenaline. Clinics (Sao Paulo). 2017 Dec;72(12):750-757. doi: 10.6061/clinics/2017(12)06. PMID 29319721
- [Result] Yin A, Yamada A, Stam WB, van Hasselt JGC, van der Graaf PH. Quantitative systems pharmacology analysis of drug combination and scaling to humans: the interaction between noradrenaline and vasopressin in vasoconstriction. Br J Pharmacol. 2018 Aug;175(16):3394-3406. doi: 10.1111/bph.14385. Epub 2018 Jul 10. PMID 29859008
- [Result] Stolk RF, van der Poll T, Angus DC, van der Hoeven JG, Pickkers P, Kox M. Potentially Inadvertent Immunomodulation: Norepinephrine Use in Sepsis. Am J Respir Crit Care Med. 2016 Sep 1;194(5):550-8. doi: 10.1164/rccm.201604-0862CP. PMID 27398737
- [Result] Hotchkiss RS, Karl IE. The pathophysiology and treatment of sepsis. N Engl J Med. 2003 Jan 9;348(2):138-50. doi: 10.1056/NEJMra021333. No abstract available. PMID 12519925
- [Result] Gordon AC, Mason AJ, Thirunavukkarasu N, Perkins GD, Cecconi M, Cepkova M, Pogson DG, Aya HD, Anjum A, Frazier GJ, Santhakumaran S, Ashby D, Brett SJ; VANISH Investigators. Effect of Early Vasopressin vs Norepinephrine on Kidney Failure in Patients With Septic Shock: The VANISH Randomized Clinical Trial. JAMA. 2016 Aug 2;316(5):509-18. doi: 10.1001/jama.2016.10485. PMID 27483065
- [Result] Smith SE, Newsome AS, Tackett RL. Prescribing of Pressor Agents in Septic Shock: A Survey of Critical Care Pharmacists. J Pharm Technol. 2019 Oct;35(5):187-193. doi: 10.1177/8755122519846164. Epub 2019 May 8. PMID 34752520
- [Result] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Result] Bauer SR, Aloi JJ, Ahrens CL, Yeh JY, Culver DA, Reddy AJ. Discontinuation of vasopressin before norepinephrine increases the incidence of hypotension in patients recovering from septic shock: a retrospective cohort study. J Crit Care. 2010 Jun;25(2):362.e7-362.e11. doi: 10.1016/j.jcrc.2009.10.005. PMID 19926252
- [Result] Hammond DA, McCain K, Painter JT, Clem OA, Cullen J, Brotherton AL, Chopra D, Meena N. Discontinuation of Vasopressin Before Norepinephrine in the Recovery Phase of Septic Shock. J Intensive Care Med. 2019 Oct;34(10):805-810. doi: 10.1177/0885066617714209. Epub 2017 Jun 15. PMID 28618919
- [Result] Bissell BD, Magee C, Moran P, Bastin MLT, Flannery AH. Hemodynamic Instability Secondary to Vasopressin Withdrawal in Septic Shock. J Intensive Care Med. 2019 Sep;34(9):761-765. doi: 10.1177/0885066617716396. Epub 2017 Jul 28. PMID 28750598
- [Result] Sacha GL, Lam SW, Duggal A, Torbic H, Reddy AJ, Bauer SR. Hypotension Risk Based on Vasoactive Agent Discontinuation Order in Patients in the Recovery Phase of Septic Shock. Pharmacotherapy. 2018 Mar;38(3):319-326. doi: 10.1002/phar.2082. Epub 2018 Feb 8. PMID 29328496
- [Result] Jeon K, Song JU, Chung CR, Yang JH, Suh GY. Incidence of hypotension according to the discontinuation order of vasopressors in the management of septic shock: a prospective randomized trial (DOVSS). Crit Care. 2018 May 21;22(1):131. doi: 10.1186/s13054-018-2034-9. PMID 29784057
- [Result] Bredhold BE, Winters SD, Callison JC Jr, Heidel RE, Allen LM, Hamilton LA. Impact of the Sequence of Norepinephrine and Vasopressin Discontinuation in Patients Recovering From Septic Shock. Hosp Pharm. 2020 Feb;55(1):26-31. doi: 10.1177/0018578718817469. Epub 2018 Dec 5. PMID 31983763
- [Result] Taylor A, Jones T, Forehand CC, Smith SE, Dykes H, Newsome AS. Vasopressor Discontinuation Order in Septic Shock With Reduced Left Ventricular Function. J Pharm Pract. 2022 Dec;35(6):879-885. doi: 10.1177/08971900211015080. Epub 2021 May 12. PMID 33977793
- [Result] Song X, Liu X, Evans KD, Frank RD, Barreto EF, Dong Y, Liu C, Gao X, Wang C, Kashani KB. The order of vasopressor discontinuation and incidence of hypotension: a retrospective cohort analysis. Sci Rep. 2021 Aug 17;11(1):16680. doi: 10.1038/s41598-021-96322-7. PMID 34404892
- [Derived] Mallmann C, Galiotto TMB, de Oliveira MS, Moraes RB. Reduction of norepinephrine versus vasopressin in the stabilization phase of septic shock: RENOVA clinical trial. Med Intensiva (Engl Ed). 2025 Oct;49(10):502147. doi: 10.1016/j.medine.2025.502147. Epub 2025 Jan 30. PMID 39890531
- See also: Borges RB, et al. Power and Sample Size for Health Researchers: uma ferramenta para cálculo de tamanho amostral e poder do teste voltado a pesquisadores da área da saúde. — http://seer.ufrgs.br/hcpa/article/view/109542